CLINICAL TRIAL: NCT03130829
Title: A Randomized, Double-blind, Placebo-controlled, Parallel, Pilot Study to Evaluate the Quality of Life Improvement of Oral Oligo Fucoidan as an Adjuvant in Subjects Receiving Platinum-based Chemotherapy With NSCLC
Brief Title: To Evaluate the QoL Improvement of Oral Oligo Fucoidan in Subjects Receiving Platinum-based Chemotherapy With NSCLC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: target population is insufficient
Sponsor: Hi-Q Marine Biotech International, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HiQ-FUCO-002
Record Dates: First submitted 2017-04-17; First posted 2017-04-27 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: NSCLC Stage IV; NSCLC, Stage III
Keywords: NSCLC; QoL; Fucoidan
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, multicenter study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oligo Fucoidan (Experimental): Oligo Fucoidan 4.4 g, sachet, oral, twice a day from Study Day -2 to End of Treatment.
  Interventions: Dietary Supplement: Oligo Fucoidan
- Placebo (Placebo Comparator): Placebo 4.4 g, sachet, oral, twice a day from Study Day -2 to End of Treatment.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oligo Fucoidan — Oral, twice daily
  Arms: Oligo Fucoidan
Dietary Supplement: Placebo — Oral, twice daily
  Arms: Placebo

SUMMARY:
Primary Objectives:

To evaluate the Quality of Life (QoL) score of adding oral Oligo Fucoidan to platinum-based chemotherapy in comparison with placebo in subjects with Non-Small Cell Lung Cancer (NSCLC).

Secondary Objectives:

To assess the progression-free survival (PFS) and objective response rate (ORR) of adding oral Oligo Fucoidan to platinum-based chemotherapy in comparison with placebo in subjects with NSCLC.

DETAILED DESCRIPTION:
This is a pilot, randomized, double-blind, multicenter study to evaluate the QoL score of Oligo Fucoidan plus platinum-based chemotherapy versus placebo plus platinum-based chemotherapy in subjects with NSCLC. Subjects will be randomized in a 1:1 ratio to receive 4.4 g BID of Oligo Fucoidan or placebo BID. Subject randomization will be stratified by NSCLC disease stage (stage III and stage IV) and platinum-based drug (cisplatin and carboplatin).

This is a two-part study. The study treatment will be planned as follow:

1. Part I (Platinum-based Treatment Phase): Oligo Fucoidan/placebo in combination with 4~6 cycles of platinum-based chemotherapy;
2. Part II (Extension Phase): Continuous Oligo Fucoidan/placebo treatment after subject completed platinum-based chemotherapy.

The total study treatment duration of investigational product from Part I to Part II will be 6 months.

Dosing of oral Oligo Fucoidan/placebo will begin on Study Day -2, 2 days prior to the start of the platinum-based chemotherapy regimen, and will continue twice a day (BID) through the following 6-months treatment period, which includes platinum-based treatment phase and extension phase, if there's no treatment interruption. All subjects will receive platinum-based IV infusion starting on Day 1 of each cycle, 3 weeks per cycle. Subjects will continue to receive Oligo Fucoidan/placebo for 6 months until develop of treatment toxicity which in the Investigator's opinion prohibits for further therapy, or until radiographic progression of disease. Subjects who experience toxicities due to chemotherapy may require a delay in the dosing schedule or a dose modification. Should a subject not receive platinum-based chemotherapy on a scheduled cycle, a rescheduled cycle will be designated when chemotherapy is reintroduced, but no more than 2 weeks delay.

The visit for subjects who have completed platinum-based treatment phase will be considered as the End of Part I Visit (end of platinum-based treatment phase). The visit for subjects who have completed 6-months treatment period (Part I & Part II) will be considered as the End of Treatment (EOT) Visit. It is preferable that EOT Visit procedures will be conducted for subjects prior to the initiation of another anticancer therapy.

Radiographic tumor assessments will be conducted at screening period, Cycle 4, End of Platinum-based Treatment Phase, and EOT. Radiographic information will be collected according to the Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.

Toxicities will be graded at each study visit according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.

Quality of life assessment as measured by the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) as well as health-related quality of life questionnaire designed by the National Health Research Institutes (NHRI), NHRI QLQ-TCM, based on traditional Chinese medicine (TCM) perspective. Both of them will be performed at Study Day -2, Day 8 of Cycle 1, Day 1 of Cycle 3 & Cycle 5, and End of Platinum-based Treatment Phase.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects must be ≥ 20 years of age, inclusive, at time of screening.
* Life expectancy > 12 weeks.
* Subject must have cytologically or histologically confirmed NSCLC. Subjects with mixed histology tumors will be eligible. If cytology is used for diagnosis, the sample must be unequivocally NSCLC.
* Subject has Stage III or IV NSCLC disease at the time of screening.
* Subject is not amenable to surgical resection or radiation with curative intent and have not received chemotherapy for their NSCLC, no matter it is new diagnosis or relapse.
* Subject is planned to receive triweekly platinum-based chemotherapy regimen prior to randomization. (Platinum dose for cisplatin is 51~80 mg/m2, or carboplatin at AUC 4~6)
* Subject must have at least 1 measurable tumor lesion, not previously irradiated, as defined by RECIST (version 1.1).
* Subject must have no history of brain metastases or evidence of CNS tumors at screening assessment..
* Subject must have an Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2.
* Subject must be able to take oral medication.
* Subject must have adequate bone marrow, renal and hepatic function as follows:

  * Absolute neutrophil count (ANC) ≥ 1,500/mm3 (1.5 × 109/L);
  * Platelets ≥ 100,000/mm3 (100 × 109/L);
  * Hemoglobin ≥ 9.0 g/dL (5.6 mmol/L);
  * Serum creatinine concentration within the normal range (according to the standard value of each hospital);
  * Hepatic function: AST and ALT ≤ 2.5 times upper limit of normal unless liver metastases are present, then AST and ALT < 5.0 times upper limit of normal; bilirubin ≤ 1.5 times upper limit of normal (subjects with Gilbert's Syndrome may have a bilirubin ≤ 3.0 times upper limit of normal).
* Female and male patients of childbearing potential and at the risk of pregnancy must agree to use at least one of highly effective contraception method throughout the study.
* Subject must be capable of understanding and complying with parameters as outlined in the protocol and able to sign inform consent.

Exclusion Criteria:

* Subject has a known hypersensitivity to Fucoidan, platinum compounds and all other drug component of current chemotherapy.
* Subject has peripheral neuropathy ≥ grade 2.
* Subject has a history of seizure within 12 months prior to study entry.
* Subject has received more or equal to third-line biomarker-targeted therapy.
* Subject has received herbal remedies for cancer treatment, non-prescription anti-cancer supplements for cancer treatment, or traditional Chinese medicine with an approved anti-cancer indication within 2 weeks prior to randomization.
* Subject is undergone or planned to receive curative radiation therapy prior to randomization and during study. (The palliative radiation therapy such as for bony lesions is allowed, but irradiate on target lesion will not be allowed.)
* Subject has clinically significant and uncontrolled major medical condition(s) including but not limited to:

  * Uncontrolled nausea/vomiting/diarrhea;
  * Active uncontrolled infection;
  * Symptomatic congestive heart failure;
  * Unstable angina pectoris or cardiac arrhythmia;
  * Psychiatric illness/social situation that would limit compliance with study requirements;
  * History of gross hemoptysis;
  * Any medical condition, which in the opinion of the Investigator, places the subject at an unacceptably high risk for toxicities.
* Subject is pregnant or lactating.
* Subject participates in study using an investigational drug within 30 days prior to screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-26 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QoL) | Day -2 to complete of Platinum-based Treatment Phase(week18)
  Comparison of the QoL score changes from Study Day -2 to End of Platinum-based Treatment Phase between Oligo Fucoidan and placebo groups in intent to treat set (ITT) via the QoL questionnaire

SECONDARY OUTCOMES:
Quality of Life (QoL) | tinumDay -2 to C1D8(week1), Cycle 3(week9), and Cycle 5(week15) of Platinum-based Treatment Phase
  Comparison of the QoL score changes from Study Day -2 to C1D8, C3D1, and C5D1 of Platinum-based Treatment Phase between Oligo Fucoidan and placebo groups in intent to treat set (ITT) via the QoL questionnaire.
Progression-Free Survival (PFS) | Screening (baseline), Cycle 4(week12), complete of Platinum-based Treatment Phase(week18), EOT(week24), and 3 months post-treatment follow up if required
  Progression-Free Survival will be evaluated according to radiographic progression per RECIST version 1.1 and survival information (death)
Objective Response Rate (ORR) | Screening (baseline), Cycle 4(week12), complete of Platinum-based Treatment Phase(week18), EOT(week24), and 3 months post-treatment follow up if required
  Objective Response Rate will be evaluated using measurements according to RECIST version 1.1
Change of Cytokines | Screening (baseline), Cycle 3 (week 9), and complete of Platinum-based Treatment Phase(week18)
  To evaluate the changes of cytokine

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Shuang Ho Hospital, New Taipei City
  - Wan-Fang Hospital, Taipei
  - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided